CLINICAL TRIAL: NCT00136084
Title: A Collaborative Trial for the Treatment of Patients With Newly Diagnosed Acute Myeloid Leukemia or Myelodysplasia
Brief Title: Treatment of Patients With Newly Diagnosed Acute Myeloid Leukemia or Myelodysplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML02; 5R01CA113482 (NIH)
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Results first posted 2010-03-26 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-11

CONDITIONS: Leukemia, Myelocytic, Acute
Keywords: Leukemia,Erythroblastic, Acute; Erythroblastic Leukemia, Acute; Leukemia, Myeloid, Acute; Myeloid Leukemia, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute | interventions — Cladribine; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Etoposide; Gemtuzumab; Asparaginase; Mercaptopurine; Methotrexate; Mitoxantrone; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HDAC (High-Dose Cytarabine) (Experimental): Since limited characters are allowed in this passage, please see detailed Description for HDAC.
  Interventions: Drug: Cladribine, Cyclophosphamide, Cytarabine, Daunorubicin, Dexamethasone
- LDAC (Low-Dose Cytarabine) (Experimental): Since limited characters are allowed in this passage, please see detailed Description for LDAC.
  Interventions: Drug: Etoposide, Cytarabine, Gemtuzumab, L-asparaginase, Mercaptopurine, methotrexate, Mitoxantrone, Prednisone, Vincristine

INTERVENTIONS:
Drug: Cladribine, Cyclophosphamide, Cytarabine, Daunorubicin, Dexamethasone — Since limited characters are allowed in this passage, please see detailed Description to know the dosage, dosage form, frequency of administration for the above mentioned drugs
  Arms: HDAC (High-Dose Cytarabine)
Drug: Etoposide, Cytarabine, Gemtuzumab, L-asparaginase, Mercaptopurine, methotrexate, Mitoxantrone, Prednisone, Vincristine — Since limited characters are allowed in this passage, please see detailed Description to know the dosage, dosage form, frequency of administration for the above mentioned drugs
  Arms: LDAC (Low-Dose Cytarabine)

SUMMARY:
The purpose of this study is to compare the effectiveness of two multi-agent chemotherapy regimens using different dosages of cytarabine to eliminate all detectable leukemia.

DETAILED DESCRIPTION:
The study compares the effectiveness of two doses of cytarabine combined with set doses of daunomycin and etoposide as an initial course of chemotherapy to eliminate minimal residual disease. Subsequent therapy is tailored according to cytogenetic risk features, assessments of minimal residual disease, and availability of a suitable donor for bone marrow transplant. Patients with higher risk disease features are given more intense therapy. For higher risk groups, transplant is given to patients with suitable donors.

Secondary objectives include:

* To assess the prognostic value of biological markers in childhood Acute Myeloid leukemia (AML).
* To compare the amounts of leukemia cells in the blood and bone marrow to study minimal residual disease(MRD).
* To relate non-invasive cardiac evaluation with health-related quality of life in AML patients treated with cardiotoxic therapy during and following therapy.

Detailed Description of Treatment Plan Induction I Patients will be randomly assigned to receive induction therapy that consists of daunomycin, etoposide, and high-dose or low-dose cytarabine.

High-Dose Cytarabine (HDAC) arm:

Cytarabine 3 gm/m2 IV days 1, 3, 5 Daunomycin 50 mg/m2 IV days 2, 4, 6 Etoposide 100 mg/m2 IV days 2-6

Low-Dose Cytarabine(LDAC) arm:

Cytarabine 100 mg/m2 IV days 1-10 (20 doses) Daunomycin 50 mg/m2 IV days 2, 4, 6 Etoposide 100 mg/m2 IV days 2-6

Induction II

Patients who have < 1% MRD after Induction I will receive daunomycin, cytarabine, etoposide (ADE):

Daunomycin 50 mg/m2 IV days 1, 3, 5 Cytarabine 100 mg/m2 IV 1-8 (16 doses) Etoposide 100 mg/m2 IV days 1-5

Patients who have ≥ 1% MRD after Induction I will receive daunomycin, cytarabine, etoposide (ADE) + gemtuzumab ozogamicin:

Daunomycin 50 mg/m2 IV days 1, 3, 5 Cytarabine 100 mg/m2IV days 1-8 (16 doses) Etoposide: 100 mg/m2 IV on days 1-5 Gemtuzumab ozogamicin (GO) 3 mg/m2 IV on day 1.

Consolidation I (Chemotherapy course 3)

The chemotherapy administered in course 3 will be based on the participant's response and cytogenetic/morphologic subgroup

MRD+ patients (except those who received ADE + GO) Gemtuzumab ozogamicin 6 mg/m2 IV on day 1

MRD+ patients who had No response(NR) to induction I

These patients should proceed to Stem Cell Transplant (SCT) as soon as possible. In cases where SCT is delayed (e.g., during searches for unrelated donors), these patients should receive chemotherapy according to their cytogenetic or morphologic subtype until the time of SCT.

MRD- patients (i.e., patients who were MRD- after ADE or after GO) will receive risk-based intensification (RBI)

t(9;11) and inv(16) Cytarabine 500 mg/m2/day by continuous infusion for 120 hours Cladribine (2CDA) 9 mg/m2: IV over 30 minutes daily for 5 days

Amend 8 M4/M5 without t(9;11) or inv(16): CE Cytarabine 3 gm/m2 IV q12h x 6 doses (days 1-3) by continuous infusion for 3 hours. Etoposide 125 mg/m2 IV on days 2-5 by continuous infusion for at least one hour

t(8;21) and others: HAM Cytarabine 3 g/m2 IV x 6 doses (days 1-3) Mitoxantrone 10 mg/m2 IV days 3-4

Standard-risk patients with matched related donors and high-risk patients will proceed to stem cell transplant per institutional practice

Consolidation II (Chemotherapy course 4):

Cytarabine 3 gm/m2 IV q12 hours on days 1, 2, 8, 9 (8 doses) L-Asparaginase 6000 Units/m2 IM 3 hours after 4th and 8th doses of cytarabine

Consolidation III (Chemotherapy course 5) Mitoxantrone 10 mg/m2 IV days 1-3 Cytarabine 1 gm/m2 IV over 2 hours q12 hours on days 1-3 (6 doses)

Patients who are in first remission are eligible to be enrolled on the St. Jude protocols NKAML protocol and receive Natural Killer (NK) cell therapy instead of Consolidation III or after Consolidation III. At the discretion of their primary physician, these patients will be offered the option of enrolling on NKAML.

Some patients with biphenotypic leukemia respond poorly to AML-directed therapy, but respond quite well to lymphoid-directed therapy. Patients with such markers who have no response to induction I or who fail to achieve complete response (CR) after induction II will therefore receive lymphoid directed induction therapy. Other biphenotypic patients will continue to receive AML-directed therapy as described above

All patients will undergo lumbar puncture and receive an age-appropriate dose of intrathecal (IT) cytarabine at the time of diagnosis.

Patients without Central Nervous System disease (CNS)(i.e., less than 5 leukocytes per microliter of CSF (colony-stimulating factor) will receive one dose of intrathecal (IT) methotrexate, hydrocortisone, and cytarabine (MHA) with each course of chemotherapy beginning with induction II.

Patients with overt CNS leukemia (more or equal to 5 leukocytes per l microliter of CSF and the presence of leukemic blast cells on CSF cytospin) will receive weekly IT MHA therapy beginning 1 week after the initial dose of IT cytarabine and continuing until the CSF is free of blast cells (minimum number of doses, 4). These patients will then receive 4 additional doses of intrathecal therapy with methotrexate, hydrocortisone, and cytarabine (IT MHA) (minimum total number of doses, 8) at approximately 1-month intervals (generally given with each subsequent course of chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia by immunophenotyping, morphology, and cytochemical staining; myelodysplasia; or biphenotypic leukemia.
* Age less than or equal to 21 years at time of study entry.
* No prior therapy for this malignancy (patients with secondary AML following treatment of primary malignancy are eligible) except for one dose of intrathecal therapy.
* Negative pregnancy test
* Patient does not have Down syndrome, acute promyelocytic leukemia (APL), or juvenile myelomonocytic leukemia (JMML)

Exclusion Criteria:

* Positive pregnancy test
* Down syndrome, acute promyelocytic leukemia (APL), or juvenile myelomonocytic leukemia (JMML)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 238 (Actual)
Dates: Start 2002-08; Primary Completion 2008-07 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rubnitz, M.D., PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (8):
- United States (8):
  - Stanford University Medical Center, Palo Alto, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Michigan (Wayne State University), Detroit, Michigan
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Children's Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] Elsayed AH, Rafiee R, Cao X, Raimondi S, Downing JR, Ribeiro R, Fan Y, Gruber TA, Baker S, Klco J, Rubnitz JE, Pounds S, Lamba JK. A six-gene leukemic stem cell score identifies high risk pediatric acute myeloid leukemia. Leukemia. 2020 Mar;34(3):735-745. doi: 10.1038/s41375-019-0604-8. Epub 2019 Oct 23. PMID 31645648
- [Derived] Gamazon ER, Lamba JK, Pounds S, Stark AL, Wheeler HE, Cao X, Im HK, Mitra AK, Rubnitz JE, Ribeiro RC, Raimondi S, Campana D, Crews KR, Wong SS, Welsh M, Hulur I, Gorsic L, Hartford CM, Zhang W, Cox NJ, Dolan ME. Comprehensive genetic analysis of cytarabine sensitivity in a cell-based model identifies polymorphisms associated with outcome in AML patients. Blood. 2013 May 23;121(21):4366-76. doi: 10.1182/blood-2012-10-464149. Epub 2013 Mar 28. PMID 23538338
- [Derived] Rubnitz JE, Inaba H, Dahl G, Ribeiro RC, Bowman WP, Taub J, Pounds S, Razzouk BI, Lacayo NJ, Cao X, Meshinchi S, Degar B, Airewele G, Raimondi SC, Onciu M, Coustan-Smith E, Downing JR, Leung W, Pui CH, Campana D. Minimal residual disease-directed therapy for childhood acute myeloid leukaemia: results of the AML02 multicentre trial. Lancet Oncol. 2010 Jun;11(6):543-52. doi: 10.1016/S1470-2045(10)70090-5. Epub 2010 May 5. PMID 20451454
- See also: St. Jude Children's Research Hospital — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 238 patients were recruited between October, 2002 and June, 2008.
Pre-assignment Details: 238 patients were enrolled on the study. This report is based on results for 223 patients. 15 patients were excluded for the following reasons: 7 were switched to lymphoid-directed therapy shortly after enrollment, 6 were determined to be ineligible shortly after enrollment (wrong diagnosis), and 2 were not randomized.
Groups:
- Arm 1: (HDAC): High-dose Cytarabine (HDAC)
- Arm 2:(LDAC): Low-dose Cytarabine (LDAC)
Period: Overall Study
Arm/Group | Arm 1: (HDAC) | Arm 2:(LDAC)
Started | 109 | 114
Completed | 61 | 72
Not Completed | 48 | 42
Not completed — Death | 12 | 5
Not completed — Unacceptable toxicity | 8 | 11
Not completed — Relapse | 20 | 23
Not completed — Lost to Follow-up | 2 | 0
Not completed — No Response | 1 | 2
Not completed — Withdrawal by Subject | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: (HDAC) | Arm 2:(LDAC) | Total
Number analyzed (Participants) | 109 | 114 | 223
Age Continuous [Mean (Standard Deviation); unit: years] | 8.57 (6.08) | 8.48 (6.32) | 8.49 (6.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 48 | 98
  Male | 59 | 66 | 125

OUTCOME MEASURES:

1. Primary Outcome: Minimal Residual Disease (MRD).
Description: Detection of Minimal Residual Disease following one course of chemotherapy where positive MRD was defined as one or more leukemic cell per 1000 mononuclear bone-marrow cells (>=0.1%).
Time Frame: Day 22 MRD measurement
Population: Of the 223 randomized patients, 205 patients were included in the day 22 MRD analysis. 18 patients were not included in the day 22 MRD analysis. 5 patients had inadequate sample for MRD, 11 patients had no suitable phenotype to determine MRD, 1 patient was not done on MRD, and 1 patient was lost for follow-up.
Measure: Number; unit: participants
Arm/Group | Arm 1: (HDAC) | Arm 2:(LDAC)
Number analyzed (Participants) | 99 | 106
participants
  MRD Positive | 31 | 43
  MRD Negative | 68 | 63
Statistical Analysis 1: Comparison: Arm 1: (HDAC) vs Arm 2:(LDAC); The study was designed to test the null hypothesis that HDAC and LDAC result in the same proportion of patients with positive MRD after 22 days. Power calculations indicate that enrollment of a total of 186 MRD-evaluable patients in a 5-stage O'Brien-Fleming group sequential design gives 80% power at the 5% level to detect a change in the MRD-positive proportion from 0.50 to 0.30. The design was developed using East statistical software; Test type: Superiority or Other; p = .1559, Cochran-Mantel-Haenszel — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.041 so that the overall level of the study is maintained at 0.05 across the 4 interim analyses and the final analysis; The p-value was computed using a Monte Carlo approximation (10000 permutations) to an exact, risk-group stratified, test; Odds Ratio (OR) = 1.624, 95% CI [.832 to 3.205] — The odds ratio is defined as the ratio of the odds that a LDAC patient is MRD positive to the odds that a HDAC patient is MRD positive

2. Secondary Outcome: Proportion of Minimal Residual Disease (MRD)+ Patients Who Become MRD- After One Course of Gemtuzumab Ozogamicin (GO)
Description: To estimate the proportion of minimal residual disease (MRD)+ patients who become MRD- after one course of gemtuzumab ozogamicin (GO)
Time Frame: Consolidation I
Population: Sixteen patients received GO treatment during consolidation I. One patient with negative MRD received GO treatment, which was not consistent with the protocol definition. 15 patients were analyzed. Out of the 15 patients, 7 patients were treated on HDAC arm and 8 patients were treated on LDAC arm.
Measure: Number; unit: Participants
Groups:
- Overall: Post-GO Treatment MRD
Arm/Group | Overall
Number analyzed (Participants) | 15
Participants
  Negative | 11
  Positive | 4
Statistical Analysis 1: Comparison: Overall; Estimate of the proportion of negative minimal residual disease; Test type: Superiority or Other; Binomial proportion; Binomial proportion = .733, 95% CI [.449 to .922]

3. Secondary Outcome: Proportion of MRD Reduction After One Course of Cytarabine + Daunomycin + Etoposide (ADE) + GO
Description: To estimate proportion of patients with MRD reduction after one course of Induction II (cytarabine + daunomycin + etoposide (ADE) + GO), who had no response to first course of induction therapy.
Time Frame: Induction II
Population: Out of the 30 patients received ADE + GO treatment, one patient had inevaluable MRD prior to and after the treatment. 29 patients were analyzed. Out of the 29 patients, 10 patients were treated on HDAC arm and 19 patients were treated on LDAC arm.
Measure: Number; unit: Participants
Groups:
- Overall: Patients who have no response to one course of induction therapy
Arm/Group | Overall
Number analyzed (Participants) | 29
Participants
  Decrease | 27
  Increase or no change | 2
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; Binomial proportion; Binomial proportion = .931, 95% CI [.772 to .992]

4. Secondary Outcome: Proportion of Patients Experienced Toxicity of Cytarabine + Daunomycin + Etoposide (ADE) + GO.
Description: To estimate proportion of patients experiencing CTC Grade 3 or 4 toxicity during Induction II (Cytarabine + Daunomycin + Etoposide (ADE) + GO), who had no response to first course of induction therapy
Time Frame: Induction II
Population: 30 patients received ADE + GO during induction II and were analyzed. Out of the 30 patients, 11 patients were treated on HDAC arm, and 19 patients were treated on LDAC arm.
Measure: Number; unit: Participants
Arm/Group | Overall
Number analyzed (Participants) | 30
Participants
  Experienced Grade 3 or 4 toxicities | 27
  Did not experience Grade 3 or 4 toxicities | 3
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; Binomial proportion; Binomial proportion = .9, 95% CI [.735 to .979]

5. Secondary Outcome: To Estimate the Overall Event-free Survival (EFS) of AML Patients Who Undergo Risk-adapted and Genotype-directed Therapy
Description: Overall event-free survival (EFS) was defined as the time from study enrollment to induction failure, relapse, secondary malignancy, death, or study withdrawal for any reason, with event-free patients censored on the date of the last follow-up
Time Frame: Five Year
Population: 238 patients were enrolled on the study. Out of 238, 6 were determined to be ineligible and 2 were not randomized. Of the 230 patients, 14 bi-phenotypic leukemia patients were excluded. 216 AML patients were included to estimate EFS.
Measure: Number; unit: Percentage of Participants
Groups:
- Overall: Evaluation of all study participants
Arm/Group | Overall
Number analyzed (Participants) | 216
Percentage of Participants | 62.4

6. Secondary Outcome: To Assess Whether Inhibition of DNA Synthesis is Greater After High-dose Ara-C (HDAC) Than After Low-dose Ara-C (LDAC) Therapy
Description: Inhibition of DNA synthesis is defined as the percentage of DNA synthesis rate at 24-hour post-araC treatment over DNA synthesis rate pre-araC treatment.
Time Frame: Measurements were assessed in Induction I chemotherapy
Population: Of 232 eligible patients, 49 had DNA synthesis rate performed prior to araC treatment. Of the 49 patients, 23 had no 24-hr samples and 3 did not have enough cells in 24-hr samples. 21 patients with both pre and post araC samples were included in the DNA inhibition study. Of the 21 patients, 9 were treated on HDAC and 12 were treated on LDAC.
Measure: Mean (Standard Error); unit: Percent Inhibition of DNA Synthesis
Groups:
- Arm 1: (HDAC): High-dose Cytarabine (Ara-C) (HDAC)
- Arm 2:(LDAC): Low-dose Cytarabine (Ara-C) (LDAC)
Arm/Group | Arm 1: (HDAC) | Arm 2:(LDAC)
Number analyzed (Participants) | 9 | 12
Percent Inhibition of DNA Synthesis | 60.6 (16.0) | 72.8 (15.6)
Statistical Analysis 1: Comparison: Arm 1: (HDAC) vs Arm 2:(LDAC); Test type: Superiority or Other; p = 0.60, t-test, 2 sided

7. Secondary Outcome: Relationship of Inhibition of DNA Synthesis and Clinical Response
Description: Clinical response is defined as MRD (minimal residual disease) measured by flow cytometry at day 22. The MRD at day 22 is classified as positive (with MRD) or negative (no detectable MRD). The relation between inhibition of DNA synthesis and MRD was performed by logistic regression. In the model, logit of probability of MRD positive was regressed on inhibition of DNA synthesis.
Time Frame: Measurements were assessed in Induction I chemotherapy
Population: Of 232 eligible patients, 49 had DNA synthesis rate performed prior to araC treatment. Of the 49 patients, 23 had no 24-hr samples and 3 did not have enough cells in 24-hr samples. 21 patients with both pre and post araC samples were included in the DNA inhibition study. 17 of the 21 patients had evaluable day 22 MRD.
Measure: Mean (Standard Error); unit: Percent inhibition of DNA Synthesis
Groups:
- Overall: 17 of the 232 eligible patients
Arm/Group | Overall
Number analyzed (Participants) | 17
Percent inhibition of DNA Synthesis | 66.7 (12.6)
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p = 0.2287, Regression, Logistic; Odds Ratio, log = -0.0139, 95% CI 2-sided [-0.0365 to 0.00873]

ADVERSE EVENTS:
Time Frame: Adverse events have been collected from study inception (October, 2002) through February, 2009.
Arm/Group | Arm 1: (HDAC) | Arm 2:(LDAC)
Serious Adverse Events (participants affected / at risk) | 23/109 | 19/114
Other Adverse Events (participants affected / at risk) | 107/109 | 112/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: (HDAC) (N=109) | Arm 2:(LDAC) (N=114)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute vascular leak syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 5 (8) | 3 (3)
Arachnoiditis/meningismus/radiculitis (Nervous system disorders) | 1 (1) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0 (0)
CNS hemorrhage/bleeding (Nervous system disorders) | 0 (0) | 2 (4)
Cardiac left ventricular function (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular/Arrhythmia-Other (Cardiac disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
DIC (disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 1 (1) | 4 (7)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (Infections and infestations) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hallucinations (Nervous system disorders) | 0 (0) | 1 (1)
Hemorrhage-Other (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemorrhage/bleeding associated with surgery (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 6 (8) | 4 (4)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e (Infections and infestations) | 13 (19) | 10 (15)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 1 (3)
Infection without neutropenia (Infections and infestations) | 1 | 1 (1)
Infection/Febrile Neutropenia-Other (Infections and infestations) | 0 (0) | 1 (3)
Lipase (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peripheral arterial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 1 (1) | 0 (0)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 1 (1) | 0 (0)
Seizure(s) (Nervous system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Thrombosis/embolism (Cardiac disorders) | 0 (0) | 1 (1)
Typhlitis (inflammation of cecum) (Gastrointestinal disorders) | 0 (0) | 2 (2)
Veno-Occlusive Dease (VOD) (Vascular disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Wound-infectious (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: (HDAC) (N=109) | Arm 2:(LDAC) (N=114)
Abdominal pain or cramping (General disorders) | 11 (12) | 0 (0)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 6 (8) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 17 (19) | 16 (19)
Anorexia (Gastrointestinal disorders) | 23 (28) | 16 (26)
Bilirubin (Hepatobiliary disorders) | 7 (8) | 0 (0)
Colitis (Gastrointestinal disorders) | 6 (7) | 0 (0)
Conjunctivitis (Eye disorders) | 7 (7) | 0 (0)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 6 (6)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 21 (26) | 20 (27)
Epistaxis (Blood and lymphatic system disorders) | 7 (9) | 9 (14)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 69 (138) | 92 (181)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (Infections and infestations) | 0 (0) | 8 (9)
GGT (Gamma-Glutamyl transpeptidase) (Hepatobiliary disorders) | 14 (21) | 8 (9)
Gastrointestinal-Other (Gastrointestinal disorders) | 8 (8) | 0 (0)
Headache (General disorders) | 6 (7) | 9 (11)
Hemorrhage-Other (Blood and lymphatic system disorders) | 0 (0) | 12 (14)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 15 (21) | 10 (13)
Hyperkalemia (Metabolism and nutrition disorders) | 7 (8) | 6 (14)
Hypertension (Cardiac disorders) | 8 (9) | 7 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 12 (13) | 12 (17)
Hypokalemia (Metabolism and nutrition disorders) | 37 (79) | 38 (84)
Hypomagnesmia (Metabolism and nutrition disorders) | 8 (9) | 7 (11)
Hyponatremia (Metabolism and nutrition disorders) | 6 (8) | 9 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 12 (14) | 12 (14)
Hypotension (Cardiac disorders) | 11 (14) | 20 (21)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 17 (19)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e (Infections and infestations) | 83 (193) | 82 (178)
Infection without neutropenia (Infections and infestations) | 10 (10) | 13 (15)
Lipase (Metabolism and nutrition disorders) | 6 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 8 (11)
Pain-Other (General disorders) | 6 (6) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (9)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 10 (10) | 0 (0)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 18 (21) | 8 (9)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 15 (18) | 19 (22)
Typhlitis (inflammation of cecum) (Gastrointestinal disorders) | 8 (10) | 16 (17)
Vomiting (Gastrointestinal disorders) | 14 (15) | 15 (20)
Wound-infectious (Skin and subcutaneous tissue disorders) | 0 (0) | 11 (12)
Wound-non-infectious (Skin and subcutaneous tissue disorders) | 9 (10) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes